CLINICAL TRIAL: NCT04108988
Title: A Digital Intervention for HIV Prevention in Black Adolescent Girls
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2000026487; 1R21HD098031-01 (NIH)
Record Dates: First submitted 2019-09-26; First posted 2019-09-30 (Actual); Results first posted 2023-11-08 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-10

CONDITIONS: HIV; Risk Reduction Behavior
Keywords: Black adolescent girls
MeSH Terms: conditions — Risk Reduction Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- InvestiDate Intervention (Experimental): One Night Stan will be adapted as a multiplayer videogame called InvestiDate based on the card game prototype with a focus on a slightly younger age group.
  Interventions: Behavioral: InvestiDate
- Non-Health Related Game (Placebo Comparator): Participants in the non-health related game group will play a multiplayer game unrelated to the content of InvestiDate.
  Interventions: Other: Non-Health Related Video Game

INTERVENTIONS:
Behavioral: InvestiDate — Participants will be randomly assigned to play either InvestiDate (n=40), or the non-health related attention and time control condition multiplayer videogame (n=40).
  Arms: InvestiDate Intervention
Other: Non-Health Related Video Game — Participants will be randomly assigned to play either InvestiDate (n=40), or the non-health related attention and time control condition multiplayer videogame (n=40).
  Arms: Non-Health Related Game

SUMMARY:
The purpose of this study is to develop and evaluate an innovative behavioral HIV prevention videogame intervention to bolster motivation and provide skill-building opportunities to improve Black adolescent girls' ability to negotiate around risk including advocating for partner HIV/sexually transmitted infection (STI) testing, increasing their knowledge and awareness of HIV/STIs, and for reducing sexual risk-taking behaviors.

DETAILED DESCRIPTION:
This study will develop and evaluate a multiplayer videogame aimed at Black adolescent girls with the intent of teaching the ability to negotiate around risk including advocating for partner HIV/STI testing, increasing their knowledge and awareness of HIV/STIs, and for reducing sexual risk-taking behaviors.

The intervention will be developed and delivered as a social, multiplayer videogame, a compelling context for Black adolescent girls who constantly interact and seek counsel from their peers. To this end, the Specific Aims, focusing on Black adolescent girls aged 14-18 years, are to:

1. (Phase 1) Translate the culturally and socially-tailored card game One Night Stan to a multiplayer videogame called InvestiDate using game design and content experts and focus group input from 30 Black adolescent girls.
2. (Phase 2) Conduct a pilot randomized controlled trial comparing the multiplayer videogame InvestiDate (the new adaptation of the One Night Stan intervention) vs. an attention/control non-health-related multiplayer videogame with 80 participants collecting assessment data at baseline, one, and four months to:

   1. Determine the intervention's acceptability and feasibility by collecting quantitative and qualitative data on Black adolescent girls' satisfaction and gameplay experience of the intervention.
   2. Determine the preliminary impact of the intervention on knowledge (information), intentions/attitudes (motivation), social norms, and behavioral skills as related to: i) HIV/STI testing and partner testing and ii) condom use, and iii) sexual risk behavior reduction, such as alcohol and drug use.

ELIGIBILITY:
Inclusion Criteria:

Both phases (includes focus groups- Phase 1)

* Black (race)
* Heterosexual
* Currently enrolled in high school

Pilot Test (Phase 2)

* Ability to participate in web-based videogame
* Willing to sit for at least 60 minutes (to play the game)
* No HIV testing in the last 12 months
* Ability to provide assent or parental/guardian consent

Exclusion Criteria:

* Failure to meet inclusion criteria

Ages: 14 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 117 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-09-24 (Actual); Study Completion 2022-09-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Hieftje, PhD, Principal Investigator — Yale University
Locations (1):
- Kimberly Hieftje, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Budge M, Opara I, Weser VU, Sands BE, Hieftje KD. Black Adolescent Females' Perceptions of PrEP for HIV Risk Reduction. J Int Assoc Provid AIDS Care. 2023 Jan-Dec;22:23259582231206934. doi: 10.1177/23259582231206934. PMID 37853731
- [Derived] Weser V, Opara I, Budge M, Duncan L, Fernandes CF, Hussett-Richardson S, Sands B, Hieftje K. Pilot-testing a Multiplayer HIV and Sexually Transmitted Infection Prevention Video Game Intervention for Black Adolescent Girls: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2023 Jan 23;12:e43666. doi: 10.2196/43666. PMID 36689272

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | InvestiDate Intervention | Non-Health Related Game
Started | 61 (61 were randomized to this arm.) | 56 (56 were randomized to this arm.)
Consent and Baseline (Excluded participants did not attend initial meeting for consenting, baseline and gameplay.) | 40 | 39
Completed Post Gameplay Survey | 40 | 38 (One participant did not attend the session.)
Completed One Month Follow-up | 40 | 39
Completed Four Month Follow-up | 38 (Two participants did not respond within the collection window.) | 39
Completed | 40 | 39
Not Completed | 21 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | InvestiDate Intervention | Non-Health Related Game | Total
Number analyzed (Participants) | 40 | 39 | 79
Age, Customized [Count of Participants; unit: Participants] — One participant turned 19 during the week that elapsed between recruitment and baseline data collection.
  Participants
    14 | 3 | 4 | 7
    15 | 7 | 3 | 10
    16 | 11 | 14 | 25
    17 | 14 | 6 | 20
    18 | 4 | 12 | 16
    19 | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 39 | 79
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 37 | 35 | 72
  Multi-Racial | 3 | 4 | 7
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 37 | 36 | 73
Region of Enrollment [Number; unit: participants]
  United States | 40 | 39 | 79
Sexual Orientation [Count of Participants; unit: Participants]
  Straight or heterosexual | 19 | 25 | 44
  Bisexual | 14 | 11 | 25
  Questioning or unsure | 5 | 3 | 8
  Queer | 1 | 0 | 1
  Asexual | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Feasibility Assessed Using Change in Retention Rates
Description: Feasibility of this intervention is assessed by the percent of total questionnaires returned out of all distributed at each time point to assess retention rates. Rates >80% indicate high retention.
Time Frame: Baseline, 1 month and 4 months
Measure: Number; unit: percentage of questionnaires returned
Arm/Group | InvestiDate Intervention | Non-Health Related Game
Number analyzed (Participants) | 40 | 39
percentage of questionnaires returned
  Baseline | 97.5 | 97.4
  1 month | 97.5 | 100
  4 months | 92.5 | 100

2. Primary Outcome: Acceptability Assessed Via Self-reported Survey
Description: Acceptability of the intervention condition is assessed via self-reported survey at the post gameplay time point using the game experience and satisfaction questionnaire, which is a 10-item scale with 4-point Likert-type responses ranging from 1 (strongly disagree) to 4 (strongly agree). Total score range 10-40. Data were collected from participants in the experimental group only. Higher scores indicate stronger agreement with the statement.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | InvestiDate Intervention
Number analyzed (Participants) | 40
score on a scale
  I would play this game again | 3.64 (0.54)
  I was frustrated with this game | 1.54 (0.56)
  I would make decisions in real life like I made them in the game | 3.44 (0.75)
  I liked the way the game looked | 3.51 (0.68)
  I felt connected to the characters in the game | 3.03 (0.67)
  I felt responsible for the choices I made in the game | 3.54 (0.51)
  I liked talking with other players about what was happening in the game | 3.51 (0.56)
  I enjoyed playing the game agree | 3.75 (0.44)
  The game was challenging | 1.97 (0.81)
  I would tell my friends to play this game | 3.44 (0.64)

3. Primary Outcome: Acceptability Assessed by Favorite Investidate Activities
Description: Participants were asked to indicate (from a list) their favorite activity in the game. The data presented here indicates the total number of participants in the experimental group that selected each activity as their favorite.
Time Frame: Month 4
Measure: Count of Participants; unit: Participants
Arm/Group | InvestiDate Intervention
Number analyzed (Participants) | 39
Participants
  Investigate a guy | 21
  Trivia | 11
  Presentation | 3
  Chat with a guy | 3
  Chat with a doctor | 0
  Chat with a friend | 0
  Videos with advice from Chelsea and Brandon | 1

4. Primary Outcome: Total Time Playing
Description: The mean total time spent playing the videogame
Time Frame: Month 4
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- InvestiDate Intervention: One Night Stan will be adapted as a multiplayer videogame called InvestiDate based on the card game prototype with a focus on a slightly younger age group.
  InvestiDate: Participants will be randomly assigned to play either InvestiDate or the non-health related attention and time control condition multiplayer videogame.
Arm/Group | InvestiDate Intervention
Number analyzed (Participants) | 40
minutes | 105.56 (12.92)

5. Primary Outcome: Change From Baseline at 4 Months: HIV/STI Testing- Self
Description: HIV/STI Testing- self will be used to determine if individuals who play InvestiDate will report more HIV/STI testing and partner testing in comparison to the control condition. Investigators will conduct a longitudinal analysis using a hierarchical linear mixed models approach to compare participants in the intervention group to participants in the control group on reported participant and partner HIV/STI testing from baseline across all follow-up assessments. Data presented here shows the number of participants who said YES they had been tested out of the total number of participants in each group that responded to the question.
Time Frame: Baseline, 1 month and 4 months
Population: The data represented shows the number of participants that reported testing of the total number of participants in each group that responded to the question.
Measure: Count of Participants; unit: Participants
Arm/Group | InvestiDate Intervention | Non-Health Related Game
Number analyzed (Participants) | 40 | 39
Participants
  Baseline | 4 | 8
  1 month: number analyzed (Participants) | 38 | 38
  1 month | 2 | 9
  4 months: number analyzed (Participants) | 37 | 31
  4 months | 4 | 8
Statistical Analysis 1: Comparison: InvestiDate Intervention vs Non-Health Related Game; P value at 4 months; Test type: Superiority; p = 0.248, Chi-squared
Statistical Analysis 2: Comparison: InvestiDate Intervention vs Non-Health Related Game; P value at 1 month; Test type: Superiority; p = 0.022, Chi-squared
Statistical Analysis 3: Comparison: InvestiDate Intervention vs Non-Health Related Game; P value at baseline; Test type: Superiority; p = 0.193, Chi-squared

6. Primary Outcome: Change From Baseline at 4 Months: HIV/STI Testing- Partner
Description: HIV/STI Testing- partner will be used to test the hypothesis that individuals who play InvestiDate will report more HIV/STI testing and partner testing in comparison to the control condition. The investigators will conduct a longitudinal analysis using a hierarchical linear mixed models approach to compare participants in the intervention group to participants in the control group on reported participant and partner HIV/STI testing from baseline across all follow-up assessments.
Time Frame: Baseline, 1 month and 4 months
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | InvestiDate Intervention | Non-Health Related Game
Number analyzed (Participants) | 40 | 39
Participants
  Baseline | 8 | 10
  1 month: number analyzed (Participants) | 38 | 39
  1 month | 8 | 11
  4 months: number analyzed (Participants) | 37 | 39
  4 months | 4 | 8
Statistical Analysis 1: Comparison: InvestiDate Intervention vs Non-Health Related Game; P value at 4 months; Test type: Superiority; p = 0.246, Chi-squared
Statistical Analysis 2: Comparison: InvestiDate Intervention vs Non-Health Related Game; P value at 1 month; Test type: Superiority; p = 0.467, Chi-squared
Statistical Analysis 3: Comparison: InvestiDate Intervention vs Non-Health Related Game; P value at baseline; Test type: Superiority; p = 0.550, Chi-squared

7. Secondary Outcome: Change in Use of Condoms
Description: At each time point, participants responded to the item "Did you use a condom the last time you had sex?" Response options were "yes", "no", and "I have never had sex". Data presented here shows the number of participants who answered YES out of the number of people in each group that responded to the question.
Time Frame: Baseline, 1 month and 4 months
Population: Not all participants responded to the question at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | InvestiDate Intervention | Non-Health Related Game
Number analyzed (Participants) | 39 | 39
Participants
  Baseline | 11 | 9
  1 month: number analyzed (Participants) | 38 | 39
  1 month | 7 | 8
  4 months: number analyzed (Participants) | 37 | 39
  4 months | 4 | 7
Statistical Analysis 1: Comparison: InvestiDate Intervention vs Non-Health Related Game; P value at month 4; Test type: Superiority; p = 0.596, Chi-squared
Statistical Analysis 2: Comparison: InvestiDate Intervention vs Non-Health Related Game; P value at 1 month; Test type: Superiority; p = 0.974, Chi-squared
Statistical Analysis 3: Comparison: InvestiDate Intervention vs Non-Health Related Game; P value at baseline; Test type: Superiority; p = 0.651, Chi-squared

8. Secondary Outcome: Change in Self-Efficacy to Use Condoms (SECU) Using the Condom Use Self-Efficacy Scale (CUSES)
Description: The CUSES is a 28 item self-report questionnaire which elicits responses using a five-point Likert scale format, ranging from 'strongly disagree' to 'strongly agree'. 10 of the 28 items were administered and scores were summed for each item for each participant. Each of the responses is scored as follows: 'strongly disagree' = 0, 'disagree' = 1, 'undecided' = 2, 'agree' = 3 and 'strongly agree' = 4. The possible range of scores is 0-40, with higher scores indicating greater self-efficacy.
Time Frame: Baseline, 1 month, 4 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | InvestiDate Intervention | Non-Health Related Game
Number analyzed (Participants) | 40 | 39
score on a scale
  Baseline | 24.5 (6.35) | 27.52 (5.7)
  1 month | 29.3 (5.46) | 26.61 (5.56)
  4 months | 28.3 (6.07) | 28.09 (6.64)
Statistical Analysis 1: Comparison: InvestiDate Intervention vs Non-Health Related Game; Test for the interaction between treatment and time; Test type: Superiority; p = 0.089, ANOVA; Test for the interaction between treatment and time

9. Secondary Outcome: Change in SECU Using Sexual Risk Behavior Beliefs and Self-efficacy (SRBBS)
Description: The SRBBS measure includes 3 items (e.g., "How sure ate you that you could use a condom correctly or explain to your partner how to use a condom correctly?") measured on a scale from 1 (not sure at all) to 5 (extremely sure). For each participant a mean of the 3 items was calculated. Scores range from 1-5 with higher scores indicating higher levels of self-efficacy.
Time Frame: Baseline, 1 month, 4 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | InvestiDate Intervention | Non-Health Related Game
Number analyzed (Participants) | 40 | 39
score on a scale
  Baseline | 2.87 (0.99) | 3.02 (1.07)
  1 month | 3.71 (1.13) | 3.33 (1.09)
  4 months | 3.62 (1.06) | 3.57 (0.74)
Statistical Analysis 1: Comparison: InvestiDate Intervention vs Non-Health Related Game; Test for the interaction between treatment and time; Test type: Superiority; p = 0.095, ANOVA; Test for the interaction between treatment and time

10. Secondary Outcome: Change in Self-efficacy in Refusing Sex (SER) Using the SER Subscale of the SRBBS
Description: This subscale includes three items (e.g., "Imagine that you met someone at a party. He or she wants to have sex with you. Even though you are very attracted to each other, you're not ready to have sex. How sure are you that you could keep from having sex") rated on a scale ranging from 1 (not sure at all) to 5 (extremely sure). A mean score for the three items was calculated for each participant with score ranging from 1-5. Higher scores indicating higher levels of self-efficacy for refusing sex.
Time Frame: Baseline, 1 month and 4 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | InvestiDate Intervention | Non-Health Related Game
Number analyzed (Participants) | 40 | 39
score on a scale
  Baseline | 4.03 (0.81) | 3.98 (0.87)
  1 month | 4.4 (0.75) | 3.88 (0.94)
  4 months | 4.4 (0.83) | 4.07 (0.88)
Statistical Analysis 1: Comparison: InvestiDate Intervention vs Non-Health Related Game; Test for the interaction between treatment and time; Test type: Superiority; p = 0.136, ANOVA; Test for the interaction between treatment and time

11. Secondary Outcome: Change in Self-efficacy in Communication Using the Self-efficacy for Communication (SECM) Subscale of the SRBBS
Description: Self-efficacy for communication was assessed using the SECM subscale of the SRBBS. This subscale includes three items (e.g., "Imagine that you and your partner have been having sex but have not used condoms. You really want to start using condoms. How sure are you that you could tell that person that you want to use condoms") rated on a scale ranging from 1 (not sure at all) to 5 (extremely sure). A mean score for the three items was calculated for each participant with score ranging from 1-5. Higher scores indicating higher levels of communication.
Time Frame: Baseline, 1 month and 4 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | InvestiDate Intervention | Non-Health Related Game
Number analyzed (Participants) | 40 | 39
score on a scale
  Baseline | 4.14 (0.67) | 4.13 (0.77)
  1 month | 4.45 (0.62) | 4.06 (0.87)
  4 months | 4.37 (0.74) | 4.05 (0.87)
Statistical Analysis 1: Comparison: InvestiDate Intervention vs Non-Health Related Game; Test for the interaction between treatment and time; Test type: Superiority; p = 0.133, ANOVA; Test for the interaction between treatment and time

12. Secondary Outcome: Change in Self-efficacy for PrEP
Description: Self-Efficacy for using PrEP was assessed with a 4 item survey. Each item was measured on a scale ranging from 1 (strongly disagree) to 5 (strongly agree). A mean score for the three items was calculated for each participant with score ranging from 1-5. Higher scores indicating higher levels of self-efficacy.
Time Frame: Baseline, 1 month and 4 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | InvestiDate Intervention | Non-Health Related Game
Number analyzed (Participants) | 40 | 39
score on a scale
  Baseline | 4.16 (0.78) | 4.13 (0.75)
  1 month | 4.51 (0.57) | 4.16 (0.71)
  4 months | 4.42 (0.82) | 4.32 (0.69)
Statistical Analysis 1: Comparison: InvestiDate Intervention vs Non-Health Related Game; Test for the interaction between treatment and time; Test type: Superiority; p = 0.210, ANOVA; Test for the interaction between treatment and time

13. Secondary Outcome: Change in Attitudes About Condom Use (ACU) Assessed Using the ACU Subscale of the SRBBS
Description: Attitudes about condom use were assessed using the ACU subscale of the SRBBS. This subscale includes three items scored from -2 (strongly disagree) to +2 (strongly agree). A mean score was calculated for each participant with negative mean scores indicating negative (unhealthy) attitudes about condom use and positive scores indicating positive (healthy) attitudes about condom use.
Time Frame: Baseline, 1 month and 4 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | InvestiDate Intervention | Non-Health Related Game
Number analyzed (Participants) | 40 | 39
score on a scale
  Baseline | 1.64 (0.54) | 1.57 (0.75)
  1 month | 1.72 (0.56) | 1.54 (0.71)
  4 months | 1.56 (0.67) | 1.61 (0.61)
Statistical Analysis 1: Comparison: InvestiDate Intervention vs Non-Health Related Game; Test for the interaction between treatment and time; Test type: Superiority; p = 0.392, ANOVA; Test for the interaction between treatment and time

14. Secondary Outcome: Change in Attitudes About Sexual Intercourse (ASI) Were Assessed Using the ASI Subscale of the SRBBS
Description: Attitudes about sexual intercourse were assessed using the ASI subscale of the SRBBS. This subscale includes three items scored from -2 (strongly disagree) to +2 (strongly agree). A mean score was calculated for each participant with negative mean scores indicating negative (unhealthy) attitudes about condom use and positive scores indicating positive (healthy) attitudes about sexual intercourse.
Time Frame: Baseline, 1 month and 4 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | InvestiDate Intervention | Non-Health Related Game
Number analyzed (Participants) | 40 | 39
score on a scale
  Baseline | -0.05 (0.43) | -0.06 (0.57)
  1 month | 0.09 (0.50) | 0.08 (0.58)
  4 months | -0.05 (0.51) | 0.11 (0.51)
Statistical Analysis 1: Comparison: InvestiDate Intervention vs Non-Health Related Game; Test for the interaction between treatment and time; Test type: Superiority; p = 0.411, ANOVA; Test for the interaction between treatment and time

15. Secondary Outcome: Change in Intentions to Find a Clinic to Speak to a Doctor About PrEP
Description: Intentions were measured with one item ("I intend to find a clinic in my community where I can speak to a doctor or health care provider about PrEP"). A mean score for the three items was calculated for each participant with score ranging from 1-5. Higher scores indicating stronger intentions.
Time Frame: Baseline, 1 months and 4 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | InvestiDate Intervention | Non-Health Related Game
Number analyzed (Participants) | 40 | 39
score on a scale
  Baseline | 2.58 (0.81) | 2.58 (0.89)
  1 month | 3.22 (1.15) | 3.08 (1.19)
  4 months | 3.06 (1.29) | 3.34 (1.05)
Statistical Analysis 1: Comparison: InvestiDate Intervention vs Non-Health Related Game; Test for the interaction between treatment and time; Test type: Superiority; p = 0.294, ANOVA; Test for the interaction between treatment and time

16. Secondary Outcome: Change in Sexually Transmitted Infections (STI)/HIV Knowledge
Description: STI/HIV knowledge was assessed using 12 questions for which participants could answer "true", "false", or "not sure". The answers were recoded as correct or incorrect, with "not sure" being coded as incorrect, and a sum was calculated for each participant. Scores range from 0 - 12 with higher scores indicating more STI-HIV knowledge.
Time Frame: Baseline, 1 months and 4 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | InvestiDate Intervention | Non-Health Related Game
Number analyzed (Participants) | 40 | 39
score on a scale
  Baseline | 7.76 (2.36) | 8.41 (2.05)
  1 month | 9.06 (1.59) | 8.73 (1.59)
  4 months | 9.06 (1.5) | 8.43 (1.92)
Statistical Analysis 1: Comparison: InvestiDate Intervention vs Non-Health Related Game; Test for the interaction between treatment and time; Test type: Superiority; p = 0.031, ANOVA; Test for the interaction between treatment and time

17. Secondary Outcome: Change in Norms About Condom Use (NCU) Assessed Using the NCU Subscale of the SRBBS
Description: Norms about condom use were assessed using the NCU subscale of the SRBBS. This subscale includes three items scored from -2 (strongly disagree) to +2 (strongly agree). A mean score was calculated for each participant with negative mean scores indicating negative (unhealthy) perceived about condom use and positive scores indicating positive (healthy) perceived norms about sexual intercourse.
Time Frame: Baseline, 1 months and 4 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | InvestiDate Intervention | Non-Health Related Game
Number analyzed (Participants) | 40 | 39
score on a scale
  Baseline | 0.93 (1.07) | 0.98 (0.88)
  1 month | 1.29 (0.99) | 1.03 (0.98)
  4 months | 1.17 (0.96) | 1.05 (0.91)
Statistical Analysis 1: Comparison: InvestiDate Intervention vs Non-Health Related Game; Test of interaction with treatment and time; Test type: Superiority; p = 0.262, ANOVA; Test for the interaction between treatment and time

18. Secondary Outcome: Change in Norms About Intercourse (NSI) Assessed Using the NSI Subscale of the SRBBS
Description: Norms about sexual intercourse were assessed using the NSI subscale of the SRBBS. This subscale includes three items scored from -2 (strongly disagree) to +2 (strongly agree). A mean score was calculated for each participant with negative mean scores indicating negative (unhealthy) perceived about condom use and positive scores indicating positive (healthy) perceived norms about sexual intercourse.
Time Frame: Baseline, 1 months and 4 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | InvestiDate Intervention | Non-Health Related Game
Number analyzed (Participants) | 40 | 39
score on a scale
  Baseline | 0.05 (0.54) | 0.01 (0.47)
  1 month | 0.19 (0.54) | 0.22 (0.73)
  4 months | -0.04 (0.54) | 0.25 (0.53)
Statistical Analysis 1: Comparison: InvestiDate Intervention vs Non-Health Related Game; Test for the interaction between treatment and time; Test type: Superiority; p = 0.116, ANOVA; Test for the interaction between treatment and time

19. Secondary Outcome: Change in Perceived Norms About PrEP
Description: Perceived norms about the use of PrEP were assessed using a 2 item survey. Both items were rated from 1 (not at all) to 4 (a lot). A mean of the two items was calculated for each participant with score ranging from 1-4. Higher scores indicate more positive perceived norms about the use of PrEP.
Time Frame: Baseline, 1 months and 4 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | InvestiDate Intervention | Non-Health Related Game
Number analyzed (Participants) | 40 | 39
score on a scale
  Baseline | 3.21 (0.68) | 3.08 (0.82)
  1 month | 3.33 (0.71) | 3.51 (0.54)
  4 months | 3.33 (0.64) | 3.42 (0.56)
Statistical Analysis 1: Comparison: InvestiDate Intervention vs Non-Health Related Game; Test for the interaction between treatment and time; Test type: Superiority; p = 0.016, ANOVA; Test for the interaction between treatment and time

20. Secondary Outcome: Change in Barriers to Condom Use (BCU) Assessed Using the BCU Subscale of the SRBBS
Description: The BCU subscale includes six items assessed on a scale ranging from 1 (strongly disagree) to 5 (strongly agree). A mean score was calculated for each participant with score ranging from 1-5. Higher scores indicating more perceived barriers to condom use.
Time Frame: Baseline, 1 months and 4 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | InvestiDate Intervention | Non-Health Related Game
Number analyzed (Participants) | 40 | 39
score on a scale
  Baseline | 2.53 (0.77) | 2.59 (0.86)
  1 month | 2.32 (0.87) | 2.49 (0.84)
  4 months | 2.33 (0.74) | 2.37 (0.77)
Statistical Analysis 1: Comparison: InvestiDate Intervention vs Non-Health Related Game; Test for the interaction between treatment and time; Test type: Superiority; p = 0.667, ANOVA; Test for the interaction between treatment and time

21. Secondary Outcome: Change in Behavior of Purchasing Condoms
Description: Participants reported on whether they had purchased condoms ever (baseline) or since they first played the videogame over zoom as part of this research study (1 month, 4 months). The response options were "yes" or "no". Data presented here shows the number of participants who answered YES out of the number of people in each group that responded to the question.
Time Frame: Baseline, 1 month and 4 months
Population: Data was analyzed from all participants that responded to the question at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | InvestiDate Intervention | Non-Health Related Game
Number analyzed (Participants) | 50 | 39
Participants
  Baseline | 5 | 5
  1 month: number analyzed (Participants) | 38 | 39
  1 month | 7 | 6
  4 months: number analyzed (Participants) | 37 | 39
  4 months | 2 | 7
Statistical Analysis 1: Comparison: InvestiDate Intervention vs Non-Health Related Game; P value at month 4; Test type: Superiority; p = 0.09, Chi-squared
Statistical Analysis 2: Comparison: InvestiDate Intervention vs Non-Health Related Game; P value 1 month; Test type: Superiority; p = 0.72, Chi-squared
Statistical Analysis 3: Comparison: InvestiDate Intervention vs Non-Health Related Game; P value at baseline; Test type: Superiority; p = 0.97, Chi-squared

22. Secondary Outcome: Change in Behavior of Having Looked up a Place to Get HIV or STI Testing
Description: Participants reported on whether they had looked up a place to get HIV or STI testing ever (baseline) or since they first played the videogame over zoom as part of this research study (1 month, 4 months). The response options were "yes" or "no". Data presented here shows the number of participants who answered YES out of the number of people in each group that responded to the question.
Time Frame: Baseline, 1 month and 4 months
Population: Data was analyzed from all participants that responded to the question at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | InvestiDate Intervention | Non-Health Related Game
Number analyzed (Participants) | 40 | 39
Participants
  Baseline | 8 | 16
  1 month: number analyzed (Participants) | 38 | 39
  1 month | 16 | 21
  4 months: number analyzed (Participants) | 37 | 39
  4 months | 9 | 12
Statistical Analysis 1: Comparison: InvestiDate Intervention vs Non-Health Related Game; P value at month 4; Test type: Superiority; p = 0.53, Chi-squared
Statistical Analysis 2: Comparison: InvestiDate Intervention vs Non-Health Related Game; P value at month 1; Test type: Superiority; p = 0.303, Chi-squared
Statistical Analysis 3: Comparison: InvestiDate Intervention vs Non-Health Related Game; P value at baseline; Test type: Superiority; p = 0.042, Chi-squared

23. Secondary Outcome: Change in Behavior of Having Talked With Partner About Getting Tested for HIV or STI
Description: Participants reported on whether they had talked with a partner about getting tested for HIV or STIs ever (baseline) or since they first played the videogame over zoom as part of this research study (1 month, 4 months). The response options were "yes" or "no". Data presented here shows the number of participants who answered YES out of the number of people in each group that responded to the question.
Time Frame: Baseline, 1 month and 4 months
Population: Data was analyzed from all participants that responded to the question at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | InvestiDate Intervention | Non-Health Related Game
Number analyzed (Participants) | 40 | 39
Participants
  Baseline | 8 | 10
  1 month: number analyzed (Participants) | 39 | 39
  1 month | 8 | 11
  4 months: number analyzed (Participants) | 39 | 39
  4 months | 4 | 8
Statistical Analysis 1: Comparison: InvestiDate Intervention vs Non-Health Related Game; P value at month 4; Test type: Superiority; p = 0.246, Chi-squared
Statistical Analysis 2: Comparison: InvestiDate Intervention vs Non-Health Related Game; P value at month 1; Test type: Superiority; p = 0.467, Chi-squared
Statistical Analysis 3: Comparison: InvestiDate Intervention vs Non-Health Related Game; P value at baseline; Test type: Superiority; p = 0.55, Chi-squared

24. Secondary Outcome: Change in Birth Control Use
Description: Participants were asked to indicate if they used birth control last time they had sex. The response options were "yes", "no", and "I have never had sex". Data presented here shows the number of participants who answered YES out of the number of people in each group that responded to the question.
Time Frame: Baseline, 1 month and 4 months
Population: Data was analyzed from all participants that responded to the question at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | InvestiDate Intervention | Non-Health Related Game
Number analyzed (Participants) | 39 | 39
Participants
  Baseline | 9 | 5
  1 month: number analyzed (Participants) | 38 | 39
  1 month | 4 | 3
  4 months: number analyzed (Participants) | 37 | 39
  4 months | 5 | 5
Statistical Analysis 1: Comparison: InvestiDate Intervention vs Non-Health Related Game; P value at month 4; Test type: Superiority; p = 0.987, Chi-squared
Statistical Analysis 2: Comparison: InvestiDate Intervention vs Non-Health Related Game; P value at month 1; Test type: Superiority; p = 0.898, Chi-squared
Statistical Analysis 3: Comparison: InvestiDate Intervention vs Non-Health Related Game; P value at baseline; Test type: Superiority; p = 0.238, Chi-squared

25. Secondary Outcome: Change in Behavior Regarding Refusal to Have Sex
Description: At 1 month and 4 months, participants were asked if they had refused to have sex with a partner because he would not use a condom in the time since they first played the videogame over zoom as part of this research study. The response options were "yes" or "no".
Time Frame: 1 month and 4 months
Population: Data was analyzed from all participants that responded to the question at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | InvestiDate Intervention | Non-Health Related Game
Number analyzed (Participants) | 38 | 39
Participants
  1 month: yes | 11 | 9
  1 month: no | 27 | 30
  4 months: number analyzed (Participants) | 37 | 39
  4 months: yes | 7 | 3
  4 months: no | 30 | 36
Statistical Analysis 1: Comparison: InvestiDate Intervention vs Non-Health Related Game; P value at month 4; Test type: Superiority; p = 0.148, Chi-squared
Statistical Analysis 2: Comparison: InvestiDate Intervention vs Non-Health Related Game; P value at month 1; Test type: Superiority; p = 0.557, Chi-squared

26. Secondary Outcome: Number of Participants Refusal to Have Sex
Description: At baseline participants were asked to indicate if they had refused to have sex with a partner because he would not use a condom ever. Response options were "always", "most of the time", "about half the time", "sometimes", and "never".
Time Frame: Baseline
Population: Data was analyzed from all participants that responded to the question at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | InvestiDate Intervention | Non-Health Related Game
Number analyzed (Participants) | 38 | 38
Participants
  Always | 6 | 9
  Most of the time | 1 | 3
  Sometimes | 5 | 5
  Never | 26 | 21
Statistical Analysis 1: Comparison: InvestiDate Intervention vs Non-Health Related Game; Test type: Superiority; p = 0.653, Chi-squared

27. Secondary Outcome: Number of Participants That Asked Partner About Previous Condom Use
Description: At baseline participants were asked how often they ask their sexual partners whether or not they have used a condom in previous sexual encounters? Response options were "always", "most of the time", "about half the time", "sometimes", and "never".
Time Frame: Baseline
Population: Data was analyzed from all participants that responded to the question at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | InvestiDate Intervention | Non-Health Related Game
Number analyzed (Participants) | 38 | 37
Participants
  Always | 9 | 7
  Most of the time | 3 | 3
  Sometimes | 4 | 3
  Never | 22 | 24
Statistical Analysis 1: Comparison: InvestiDate Intervention vs Non-Health Related Game; Test type: Superiority; p = 0.977, Chi-squared

28. Secondary Outcome: Number of Times Participants Asked Partner About Previous Condom Use
Description: At 1 month and 4 months, participants were asked how many times they discussed condom use with a sexual partner since first playing the videogame on zoom as part of this research study.
Time Frame: 1 month and 4 months
Measure: Mean (Standard Deviation); unit: number of times asked partner
Arm/Group | InvestiDate Intervention | Non-Health Related Game
Number analyzed (Participants) | 40 | 39
number of times asked partner
  1 month | 1.29 (2.75) | 0.59 (1.25)
  4 months | 0.92 (2.43) | 1.13 (2.90)
Statistical Analysis 1: Comparison: InvestiDate Intervention vs Non-Health Related Game; P value at month 4; Test type: Superiority; p = 0.735, t-test, 2 sided
Statistical Analysis 2: Comparison: InvestiDate Intervention vs Non-Health Related Game; P value at month 1; Test type: Superiority; p = 0.159, t-test, 2 sided

29. Secondary Outcome: Number of Times Participants Talked to Family or Adults About HIV
Description: Participants were asked how many times they had talked with their family or other adults about HIV ever (baseline) or since they played the videogame on zoom as part of this research study (1 month, 4 months).
Time Frame: baseline, 1 month and 4 months
Measure: Mean (Standard Deviation); unit: number of times talked to family/adults
Arm/Group | InvestiDate Intervention | Non-Health Related Game
Number analyzed (Participants) | 40 | 39
number of times talked to family/adults
  baseline | 1.60 (2.62) | 6.64 (22.08)
  1 month | 3.68 (16.12) | 1.82 (3.00)
  4 months | 1.3 (6.60) | 259.95 (1600.78)
Statistical Analysis 1: Comparison: InvestiDate Intervention vs Non-Health Related Game; P value at month 4; Test type: Superiority; p = 3.19, t-test, 2 sided
Statistical Analysis 2: Comparison: InvestiDate Intervention vs Non-Health Related Game; P value at month 1; Test type: Superiority; p = 0.487, t-test, 2 sided
Statistical Analysis 3: Comparison: InvestiDate Intervention vs Non-Health Related Game; P value at baseline; Test type: Superiority; p = 0.165, t-test, 2 sided

30. Secondary Outcome: Number of Times Participants Engaged in Sexual Intercourse
Description: Participants were asked how many times they had engaged in sexual intercourse ever (baseline, post-intervention) or since playing the videogame on zoom as part of this research study (1 month, 4 months).
Time Frame: baseline, 1 month and 4 months
Measure: Mean (Standard Deviation); unit: number of times had sex
Arm/Group | InvestiDate Intervention | Non-Health Related Game
Number analyzed (Participants) | 40 | 39
number of times had sex
  baseline | 14.78 (79.26) | 6.64 (8.77)
  1 month | 1.58 (6.48) | 0.50 (0.98)
  4 months | 3.24 (16.41) | 1.26 (3.01)
Statistical Analysis 1: Comparison: InvestiDate Intervention vs Non-Health Related Game; P value at month 4; Test type: Superiority; p = 0.473, t-test, 2 sided
Statistical Analysis 2: Comparison: InvestiDate Intervention vs Non-Health Related Game; P value at month 1; Test type: Superiority; p = 0.316, t-test, 2 sided
Statistical Analysis 3: Comparison: InvestiDate Intervention vs Non-Health Related Game; P value at baseline; Test type: Superiority; p = 0.345, t-test, 2 sided

31. Secondary Outcome: Number of Times Participants Engaged in Anal Sex
Description: Participants were asked how many times they had engaged in anal sex ever (baseline) or since playing the videogame on zoom as part of this research study (1 month, 4 months).
Time Frame: baseline, 1 month and 4 months
Measure: Mean (Standard Deviation); unit: number of times had sex
Arm/Group | InvestiDate Intervention | Non-Health Related Game
Number analyzed (Participants) | 40 | 39
number of times had sex
  baseline | 0.28 (1.59) | 0.08 (0.27)
  1 month | 0.55 (3.24) | 0.03 (0.16)
  4 months | 0.03 (0.16) | 0.18 (0.60)
Statistical Analysis 1: Comparison: InvestiDate Intervention vs Non-Health Related Game; P value at month 4; Test type: Superiority; p = 0.141, t-test, 2 sided
Statistical Analysis 2: Comparison: InvestiDate Intervention vs Non-Health Related Game; P value at month 1; Test type: Superiority; p = 0.314, t-test, 2 sided
Statistical Analysis 3: Comparison: InvestiDate Intervention vs Non-Health Related Game; P value at baseline; Test type: Superiority; p = 0.444, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | InvestiDate Intervention | Non-Health Related Game
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/39
Other Adverse Events (participants affected / at risk) | 0/40 | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (4):
  • Study Protocol and Statistical Analysis Plan (2021-12-19): https://cdn.clinicaltrials.gov/large-docs/88/NCT04108988/Prot_SAP_000.pdf
  • Informed Consent Form: Compound (2021-09-30): https://cdn.clinicaltrials.gov/large-docs/88/NCT04108988/ICF_001.pdf
  • Informed Consent Form: Adolescent (2021-09-30): https://cdn.clinicaltrials.gov/large-docs/88/NCT04108988/ICF_002.pdf
  • Informed Consent Form: Parent (2021-09-30): https://cdn.clinicaltrials.gov/large-docs/88/NCT04108988/ICF_003.pdf